CLINICAL TRIAL: NCT02237183
Title: A Phase I Trial of Inhaled Iloprost for the Prevention of Lung Cancer in Former Smokers
Brief Title: Iloprost in Preventing Lung Cancer in Former Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2014-01891; NCI-2014-01891 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00035; HHSN2612201200035I; NCI2013-02-01 (Other: Northwestern University); NWU2013-02-01 (Other: DCP); N01CN00035 (NIH); P30CA060553 (NIH)
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Iloprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (iloprost QID) (Experimental): Patients receive iloprost via inhalation using a nebulizer QID for 60 days.
  Interventions: Drug: Iloprost; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (placebo QID) (Placebo Comparator): Patients receive placebo via inhalation using a nebulizer QID for 60 days.
  Interventions: Other: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (iloprost BID) (Experimental): Patients receive iloprost via inhalation using a nebulizer BID for 60 days.
  Interventions: Drug: Iloprost; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm IV (placebo BID) (Placebo Comparator): Patients receive placebo via inhalation using a nebulizer BID for 60 days.
  Interventions: Other: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Iloprost — Given via inhalation
  Other Names: Ciloprost; Iloprost Clathrate; Ventavis; ZK 36374
  Arms: Arm I (iloprost QID); Arm III (iloprost BID)
Other: Placebo Administration — Given via inhalation
  Arms: Arm II (placebo QID); Arm IV (placebo BID)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies the side effects and best dose of iloprost compared with a placebo in preventing lung cancer in former smokers. Chemoprevention is the use of drugs to keep cancer from forming or coming back. Inhaled iloprost may help prevent lung cancer from forming in patients who used to smoke and who have been found to have abnormal cells in their mucus.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicity of inhalational iloprost administered to patients daily for 2 months, given four times a day (QID).

SECONDARY OBJECTIVES:

I. To evaluate the compliance QID dosing regimens. II. To evaluate the effect on endobronchial histology. III. To evaluate the effect on expectorated sputum cytology by both standard cytologic analysis and an automated three-dimensional morphologic analysis.

IV. To evaluate the effect on endobronchial brushing and biopsy gene expression of peroxisome proliferator-activated receptor gamma (PPARgamma), glutathione S-transferase mu (GSTmu), carboxylesterase 1 (Ces1), Fos-related antigen 1 (FosL1), cytochrome p4502e1, stearoyl coA desaturase 1, tumor necrosis factor (TNF) superfamily member 9, transforming growth factor beta (TGFbeta), Jun and a 46 gene panel associated with dysplasia persistence, using Affymetrix arrays.

V. To evaluate the improvement in chronic obstructive pulmonary disease (COPD) as measured by arterial blood gas (ABG) (improved ventilation perfusion matching), pulmonary function testing, 6-minute walk distance, quality of life (St. George's respiratory questionnaire, COPD assessment test [CAT]).

VI. To evaluate whether the in vitro response of cultured airway epithelial progenitor cells to iloprost is a predictor of in vivo response in study subjects.

OUTLINE: Patients are enrolled to Cohort A to completion prior to initiation of Cohort B.

COHORT A: Patients are assigned to 1 of 2 arms.

ARM I: Patients receive iloprost via inhalation using a nebulizer QID for 60 days.

ARM II: Patients receive placebo via inhalation using a nebulizer QID for 60 days.

COHORT B: Patients are assigned to 1 of 2 arms. COHORT B DISCONTINUED AS OF 03/26/2019.

ARM III: Patients receive iloprost via inhalation using a nebulizer BID for 60 days.

ARM IV: Patients receive placebo via inhalation using a nebulizer BID for 60 days.

After completion of study treatment, patients are followed up at 90 days and then annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have either sputum cytologic atypia of mild dysplasia or greater or a history of bronchial biopsy with mild or greater dysplasia within the past 12 months
* Participants must have a smoking history of 20 pack-years or greater
* Participants must have the ability to safely undergo bronchoscopy in the judgment of the investigators
* Participants must have Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Leukocytes >= 3,000/microliter
* Platelets >= 100,000/microliter
* Total bilirubin =< 2.0 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN)
* Creatinine =< 2.0 mg/dl
* The effects of iloprost on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because prostacyclins are known to be teratogenic, women of child-bearing potential and men having intercourse with a woman of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately; Note: Women are considered to be of child-bearing potential if they are not surgically sterile or are under the age of 65 and have menstruated within the last two years
* Participants must be able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Participants must not have used any tobacco product in the past year
* Participants must not be currently receiving or have previously received thiazolidinedione treatment unless sputum atypia or endobronchial dysplasia are documented again after thiazolidinedione treatment and within 12 months of entry
* Participants must not have been treated with iloprost at any time; Note: participants on the placebo arm of previous iloprost trials are eligible, but participants on the placebo arm of cohort A of this study may not be enrolled in cohort B
* Participants must not have used any other investigation agent within the last six months
* Participants must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition of iloprost
* Participants must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that in the opinion of investigators would jeopardize patient safety of data integrity; Note: individuals who are human immunodeficiency virus (HIV) positive will not necessarily be excluded, will be considered on a case-by-case basis, but will be required to meet criteria related to patient safety and data integrity, as assessed by investigators
* Participants must not have a current or prior invasive malignancy within the past 6 months; participants may enroll prior to biopsy result report, unless there are findings at bronchoscopy suggesting an invasive malignancy; history of the following curatively treated cancers during any time prior to screening is allowed: non-melanoma skin cancer, cervical carcinoma in situ, and bladder carcinoma in situ
* Participants must not have received either chemotherapy or radiotherapy within the previous 6 months; Note: participants receiving long-term adjuvant hormonal therapy (such as tamoxifen or aromatase inhibitors for breast cancer) are allowed
* Women must not be pregnant or breastfeeding; iloprost is a prostacyclin agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with iloprost, breastfeeding should be discontinued if the mother is treated with iloprost
* As iloprost inhibits platelet function, patients must not be taking anticoagulants, with the exception of aspirin or other non-steroidal anti-inflammatory medications
* Due to risk for hypotension in patients on vasodilators or antihypertensive medications, participants must not have blood pressure < 95 mm Hg systolic

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical toxicity | Up to 90 days
  Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Descriptive statistics (mean, standard deviation [SD], median, max, min and range) will be provided for toxicity. Approximate 95% confidence intervals will be used to assess the difference between treatment groups.
Treatment compliance, measured as the fraction of prescribed inhalations actually administered | Up to 60 days
  Descriptive statistics (mean, SD, median, max, min and range) will be provided for compliance. Approximate 95% confidence intervals will be used to assess the difference between treatment groups.

SECONDARY OUTCOMES:
Response of airway histology | Up to 5 years
  Will provide descriptive statistics for the effect on endobronchial histology, with the primary parameter being worst histology at matched sites; additional outcomes will be average histology, dysplasia index and response, as described.
Serum protein profiling | Up to 60 days
  Will provide descriptive statistics for the effect on serum proteins as quantitated by aptamer based analysis.
Endobronchial brushing gene expression | Up to 60 days
  Will provide descriptive statistics for the effect on endobronchial brushing gene expression, focusing on prostacyclin-targeted pathways.
Gene expression of dysplastic lesions | Up to 60 days
  Will provide descriptive statistics.
Improvement in chronic obstructive pulmonary disease (COPD) | Up to 60 days
  Will provide descriptive statistics for the improvement in COPD as measured by arterial blood gas (improved ventilation perfusion matching), pulmonary function testing, 6-minute walk distance, and quality of life (St. George's respiratory questionnaire, COPD assessment test).
Whether the in vitro response of cultured airway epithelial progenitor cells to iloprost is a predictor of in vivo response in study subjects | Up to 60 days
  Bronchial biopsies will be taken from an area suspicious for dysplasia and an area that appears normal. These will be cultured as described and transferred to an air liquid interface culture in which dysplasia is recapitulated. Cultures will be treated with either vehicle or iloprost and assessed for both self-renewal and differentiation to ciliated and secretory cells.

CONTACTS AND LOCATIONS:
Overall Officials: York E Miller, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - University of Colorado, Denver, Colorado

REFERENCES:
- [Derived] Miller YE, Ghosh M, Merrick DT, Kubala B, Szabo E, Bengtson L, Kocherginsky M, Helenowski IB, Benante K, Schering T, Kim J, Kim H, Ha D, Bergan RC, Khan SA, Keith RL. Phase Ib trial of inhaled iloprost for the prevention of lung cancer with predictive and response biomarker assessment. Front Oncol. 2023 Aug 30;13:1204726. doi: 10.3389/fonc.2023.1204726. eCollection 2023. PMID 37711198

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT02237183/Prot_SAP_000.pdf